CLINICAL TRIAL: NCT06185244
Title: Efficacy and Cost Effectiveness of Internet-delivered Trauma-focused CBT for Young People With PTSD
Brief Title: Efficacy of Internet-delivered Trauma-focused CBT for Young People With PTSD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Child and Adolescent Psychiatry, Stockholm (Industry); Save the Children (Other)
Responsible Party: Principal Investigator, Maria Bragesjo, PhD, clinical psychologist, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2023-06501-01
Record Dates: First submitted 2023-12-14; First posted 2023-12-29 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: Posttraumatic Stress Disorder
Keywords: PTSD; digital treatment; trauma-focused CBT; therapist-guided
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Outcomes Assessor
Masking Description: Blinded assessors will be used.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Therapist-supported internet delivered trauma-focused CBT (Experimental): Therapist-supported internet delivered trauma-focused CBT. The protocol mirrors the exact content of first-line treatment for children with PTSD but is delivered through a digital platform and will comprise of text-based material as well as audio files and video illustrations in an age-appropriate manner that the participant gains access to sequentially. iTF-CBT will be therapist-assisted, and each participant will have a designated therapist to guide them through treatment. Treatment will span over 12 weeks and integrates cognitive, behavioral, interpersonal, and family therapy principles as well as trauma interventions. Parallel to the child's treatment, the caregivers are provided the same components and parenting practices, and joint child-parent activities are included. Participants will have access to a therapist that will guide them through treatment in a text based format.
  Interventions: Behavioral: Therapist-supported internet-delivered trauma-focused CBT
- Therapist-supported psychoeducation and stress management (Active Comparator): Therapist-supported CBT internet-delivered treatment comprising psychoeducation about PTSD, relaxation/stress management techniques and relapse prevention. The treatment will be delivered in a digital platform for twelve weeks. Participants will have access to a therapist that will guide them through treatment in a text-based material as well as audio files and video illustrations in an age-appropriate manner that the participant gains access to sequentially.
  Interventions: Behavioral: 12 weeks of therapist-supported internet-delivered psychoeducation and stress management/relaxation for both the youth and the care giver.

INTERVENTIONS:
Behavioral: Therapist-supported internet-delivered trauma-focused CBT — 12 weeks of therapist-supported internet-delivered trauma-focused CBT for both the youth and the care giver.
  Arms: Therapist-supported internet delivered trauma-focused CBT
Behavioral: 12 weeks of therapist-supported internet-delivered psychoeducation and stress management/relaxation for both the youth and the care giver. — 12 weeks of therapist-supported internet-delivered psychoeducation and stress management/relaxation for both the youth and the care giver.
  Arms: Therapist-supported psychoeducation and stress management

SUMMARY:
The goal of this clinical trial is to compare therapist-guided internet delivered trauma-focused cognitive behavior therapy (CBT) to an active control condition comprising therapist-guided internet delivered cognitive behavioral therapy containing relaxation techniques and psychoeducation for young people with post-traumatic stress disorder regarding efficacy and cost effectiveness.

Young people with post-traumatic stress disorder will be randomly assigned to receive either 12 weeks of therapist-guided internet delivered trauma-focused cognitive behavior therapy (iTF-CBT) or therapist-guided internet delivered cognitive-behavioral therapy containing relaxation and psychoeducation.

DETAILED DESCRIPTION:
There is an urgent need for evidence-based treatments for children with PTSD that can easily be made available to a large number of afflicted. The overall aim of the project is to increase the availability of evidence-based psychological treatments for adolescents with PTSD by developing and evaluating iTF-CBT for this target group. The main objectives are to establish the efficacy, cost-effectiveness, and long-term effects of iTF-CBT for adolescents with PTSD in an RCT (N=140) by comparing guided iTF-CBT with an attention control group consisting of therapist-supported internet-delivered psychoeducation and support.

The study is a single-blind, parallel-group superiority randomized controlled trial with 240 patients (120 per arm) that will compare therapist-guided internet delivered trauma-focused cognitive behavior CBT with therapist-guided internet delivered cognitive-behavioral therapy comprising relaxation and psychoeducation. The primary outcome is the blind-rater administered Clinician-Administered PTSD Scale for DSM-5 (CAPS-5-CA). An internal pilot is built in in the design and the first 20 enrolled participants will not be randomized but receive the active intervention. They will also be asked to participate in qualitative interviews about their experience of the intervention.

Secondary outcomes are cost effectiveness, predictors of clinically meaningful change in symptoms, mediators of change, dropout rate, and negative effects.

Research questions:

1. Is guided iTF-CBT more efficacious than an active control condition (therapist-supported internet-delivered psychoeducation and support) in regard to reduction of blinded assessor rated PTSD symptom severity 1-month post-treatment?
2. Is guided iTF-CBT more cost-effective than an active control condition (therapist-supported internet-delivered psychoeducation and support) in regard to reduction of blinded assessor rated PTSD symptom severity 1-month post-treatment?
3. Are the therapeutic gains of iTF-CBT maintained at long term follow up (6 and 12 months after treatment)?
4. How do children, parents and therapists perceive iTF-CBT?

ELIGIBILITY:
Inclusion Criteria:

* 13-17 years,
* Primary PTSD diagnosis
* Fluent in Swedish
* Access to the Internet at home or can use vouchers for internet-access to their phone.
* Parent/guardian willing and able to take part in treatment.

Exclusion Criteria:

* PTSD is not the primary concern
* Initiation or adjustment of any psychotropic medication within the last 4 weeks prior to commencement of treatment
* Serious mental health symptoms, such as mania, psychosis, alcohol, or substance use disorders or current suicide risk warranting immediate clinical attention.
* Ongoing trauma-focused CBT or Eye movement desensitization and reprocessing Therapy
* Ongoing trauma-related threat

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 240 (Estimated)
Dates: Start 2024-03-11 (Actual); Primary Completion 2027-01-04 (Estimated); Study Completion 2028-01-04 (Estimated)

PRIMARY OUTCOMES:
Change in PTSD symptoms as assessed by the Clinician Administered PTSD Scale Children and Adolescent version 5 (CAPS-5-CA) | Baseline, 1-month (primary endpoint), 6-month and 12-month after treatment completion
  The CAPS-5-CA is a structured interview that assesses the Diagnostic and Statistical Manual of Mental Disorders version 5 (DSM-5) criteria for PTSD (Weathers et al., 2013). Each item is rated on a severity scale ranging from 0 (Absent) to 4 (Extreme/incapacitating) and combines information about frequency and intensity for each of the 20 symptoms. Total Score (Range 0-80 with higher scores representing more PTSD symptoms.

SECONDARY OUTCOMES:
Change in self-rated symptoms of PTSD and complex PTSD measured by The Child and Adolescent Trauma Screen (CATS-2) | Baseline, through the treatment period up to 12 weeks and 1-month, 6-month and 12-month after treatment completion
  The CATS-2 measures potentially traumatic events (PTEs), posttraumatic stress symptoms (PTSS) and impairment according to DSM-5 and ICD-11 criteria in children and adolescent from 7 to 17 years. In addition to a self-report measure for children and adolescents, the CATS-2 includes a parallel caregiver version. Posttraumatic stress symptoms in the last four weeks are then assessed using 25 items rated on a 4-point. The 25 items map directly onto the diagnostic criteria for PTSD in DSM-5 and ICD-11 PTSD and CPTSD. The DSM-5 PTSD severity score is the sum of items 1-20 (range 0-60), including only the highest score of items 9, 10, 15. The ICD-11 PTSD severity score (range 0-18) is the sum of items 2, 3, 6, 7, 17, 18. The ICD-11 CPTSD score (range 0-36) is the sum of ICD-11 PTSD severity score (2, 3, 6, 7, 17, 18) plus the sum of the ICD-11 DSO severity score (9b, 9d, 10a, 13, 14, 15a). Higher scores represents more PTSD symptoms.
Change in self-rated symptoms of depression as measured by Mood and Feelings Questionnaire (MFQ) | Baseline, immediately after treatment completion, and 1-month, 6-month and 12-month after treatment completion
  The MFQ consists of a series of 33 descriptive phrases regarding how the subject has been feeling or acting recently. Respondents are asked whether descriptions in the questionnaire are 'true', 'sometimes true' or 'not true' for them over the past two weeks. The MFQ is scored by summing together the point values of responses for each item. The response choices and their designated point values are as follows: "not true" = 0 points, "sometimes true" = 1 point, "true" = 2 points. Higher scores on the MFQ suggest more severe depressive symptoms.
Change in psychosocial impairment measured by The Education, Work and Social Adjustment Scale, Youth and Parent (EWSAS) | Baseline, immediately after treatment completion, and 1-month, 6-month and 12-month after treatment completion
  EWSAS is a short, self-reported instrument consisting of five items about psychosocial impairments rated on a nine-point Likert scale. A higher score means more severe impairment.
Change in Treatment Inventory of Costs in Psychiatric Patients (TIC-P) | Baseline, immediately after treatment completion, and 1-month, 6-month and 12-month after treatment completion
  Self-rated questionnaire on healthcare utilization and productivity losses in patients with a psychiatric disorder. The TIC-P questionnaire measures costs in two dimensions: use of health resources and loss of productivity. Lower cost is better.
Adverse events related to treatment measured by the Negative effects questionnaire | Immediately after treatment completion, 1-month, 6-month and 12-month after treatment completion
  Self-rated questionnaire on negative effects. It contains 32 items that are scored on a five point Likert-scale (0-4) and differentiates between negative effects that are attributed to treatment and those possibly caused by other circumstances. The total score of the NEQ ranges from 0 to 80 points, a higher score reflects more negative effects.
Quality of life measured by Assessment of Quality of Life KIDSCREEN-10 | Immediately after treatment completion, 1-month, 6-month and 12-month after treatment completion
  Change in subjective psychological, mental and social well-being from baseline to immediately after treatment and follow up . a higher score reflects higher health-related quality of life.
Participants satisfaction with treatment, assessed by The Client Satisfaction Questionnaire (CSQ-8). | Immediately after treatment completion.
  The CSQ-8 yields a single score measuring a single dimension of overall satisfaction. An "overall score" is calculated by summing the score on each of the eight scale item. Scores range from 8 to 32, with higher values indicating higher satisfaction.
Number of completed treatment modules | Baseline up to 12 weeks
  Data will be gathered on total number of completed modules during the 12 week treatment.
Number of messages sent and received in the digital platform | Baseline up to 12 weeks
  Data will be gathered on total number of messages sent and received back and forth between the participant and the therapist during the 12 week treatment.
Number of home work assignments made by the participant during the treatment period | up to 12 weeks
  umber of home work assignments made by the participant during the treatment period
The proportion of participants that conducts the weekly measures and further assessment points | up to the 6 months follow up
  The proportion of participants that conducts the weekly measures and further assessment points
The proportion of participants that go through the entire treatment period | up to 12 weeks
  The proportion of participants that go through the entire treatment period
Number of drop-outs from treatment | up to 12 weeks
  Number of drop-outs from treatment
Participants experience/satisfaction with treatment and assessment procedures through qualitative interviews | up to the 6-month follow up
  Participants experience/satisfaction with treatment and assessment procedures through qualitative interviews

OTHER OUTCOMES:
Differences in treatment credibility between arms | After completion of the first treatment module (week 1 from baseline)
  Measures treatment expectancy and rationale credibility. The CEQ is a 5-item measure of the treatment's credibility and the patients' expectations. The patients assess each domain on a 11-point likert scale (scored 0-10), with a total score ranging between 0-50 where higher score indicates higher credibility and higher expectations.
Differences in experience of working alliance between arms | After completion of the third module (week 3 from baseline)
  Measures the therapeutic alliance in therapy. The WAI-SR is a 12-item measure of the patient's experience of their working alliance with the therapist. The patients assess each item on a 7-point likert scale (scored 0-6), with a total score ranging between 0-72 where higher score indicates higher better working alliance according to the patient.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Bragesjö, PhD, Principal Investigator — Karolinska Institutet/Region Stockholm
Locations (1):
- Barn och ungdomspsykiatrin, BUP Internetenhet and Save the Children, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No